CLINICAL TRIAL: NCT01867892
Title: A Phase II Randomized Study of Induction Chemotherapy Followed by Concurrent Chemo-radiotherapy in Locally Advanced Pancreatic Cancer
Brief Title: A Phase II Study of Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T2212
Record Dates: First submitted 2013-05-07; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Pancreatic Cancer
Keywords: Locally Advanced Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICT of oxaliplatin,irinotecan,5-FU and leucovorinon and CCRT (Experimental): Arm1:oxaliplatin,irinotecan,5-FU and leucovorinon D1,15 every 28days for 3 cycles,RT 5,040cGy in 28 fractions/5.5 wks and 5FU 450mg/m2 iv 30min weekly
  Interventions: Drug: ICT of oxapliplatin, irinotecan, leucovorin, and fluorouracil and CCRT
- ICT of gemcitabine,oxaliplatin,5-FU,leucovorin and CCRT (Active Comparator): Arm 2:gemcitabine,oxaliplatin,5-FU,leucovorin on D1,15 every 28 days for 3 cycles,Evaluation of Tumor Response,CR/PR/SD or localized disease RT 5,040cGy in 28 fractions/ 5.5 wks Arm 2: Gem 400mg/m2 iv 40min weekly
  Interventions: Drug: ICT of Gemcitabine,oxapliplatin, leucovorin, and fluorouracil + CCRT

INTERVENTIONS:
Drug: ICT of oxapliplatin, irinotecan, leucovorin, and fluorouracil and CCRT — oxapliplatin ,irinotecan ,5FU +leucovorin ,RT 5,040cGy in 28 fractions/5.5 wks and 5FU 450mg/m2 iv 30min weekly
  Other Names: ICT of oxapliplatin,irinotecan,leucovorin,and fluorouracil and CCRT
  Arms: ICT of oxaliplatin,irinotecan,5-FU and leucovorinon and CCRT
Drug: ICT of Gemcitabine,oxapliplatin, leucovorin, and fluorouracil + CCRT — Gem ,Oxa ,5FU +LV ,RT 5,040cGy in 28 fractions/5.5 wks and Gem 400mg/m2 iv 40min weekly
  Other Names: ICT of Gemcitabine,oxapliplatin, leucovorin, and fluorouracil +CCRT
  Arms: ICT of gemcitabine,oxaliplatin,5-FU,leucovorin and CCRT

SUMMARY:
The primary end point is to evaluate the 9-month progression free survival rate and safety profile after FOLFIRINOX versus GOFL induction chemotherapy followed by concurrent chemoradiotherapy in locally advanced pancreatic cancer.

The secondary end points are to evaluate the disease control rate, overall survival time, toxicity profile and compliance after induction chemotherapy and concurrent chemoradiotherapy as well as the disease control rate after inductional chemotherapy alone in locally advanced pancreatic cancer. Translational research including pharmacogenomic study and biomarker study will also be done concomitantly.

DETAILED DESCRIPTION:
Patients should be randomized to two study arms stratified by resectability status (borderline resectable and unresectable) after enrollment. Eligible patients will be randomly assigned on a 1:1 basis to either of two study groups, using a central randomization procedure with stratification according to NCCN criteria of resectability.

After randomization, induction chemotherapy (ICT) will be administered for 3 cycles (3 months). Patients who have radiological evidence of distant dissemination will be shifted to salvage chemotherapy. Patients who have responsive, stable disease as well as those with localized progressive disease after ICT will receive concurrent chemoradiotherapy (CCRT) 3-4 weeks after the last dose of ICT. Surgical evaluation will be performed 4-6 weeks after the completion of CCRT. Patients who have respectable disease will undergo surgical resection. Postoperative adjuvant chemotherapy for 3 cycles (3 months) will be given for those who are considered to have curative resection. Patients who still have unresectable disease or non-curative resection will receive systemic chemotherapy till disease progression or unacceptable toxicity.

For Arm 1, ICT with FOLFIRINOX ( oxaliplatin 85mg/m2 for 2 hr, irinotecan 180mg/m2 for 90 min and 5FU 3000mg/m2 + LV 150mg/m2 continuous infusion 48 hr) will be administered biweekly. For Arm 2, ICT with GOFL ( 800mg/m2 gemcitabine at a fixed rate of 10mg/m2/min followed by a 2-hour oxaliplatin 85mg/m2 and then a 48-hour 3000mg/m2 5-FU and 150 mg/m2 leucovorin on day 1 and 15 every 28 days/cycle) will be given biweekly.

After three 3 cycles of ICT, patients without distant metastasis will be given CCRT with 5-FU 450mg/m2 in Arm 1, gemcitabine 400mg/m2 in Arm 2, 2 hrs before RT on day1,8,15,22,29,36. Radiation will be given 180cGy per day, 5 days a week for 28 fractions to totally 5040cGy.

If complete surgical resection is feasible, optimal surgery will be performed 4-6 weeks after CCRT. If complete surgical resection is impossible, biopsy with or without bypass surgery may be performed. Patients who have curative surgical resection will receive additional 6 cycles ( 6 months) of adjuvant chemotherapy ( Arm1, FOLFIRINOX, Arm 2, GOFL) within 4 weeks after surgery and then followed up until tumor progression. Patients who are not feasible for curative resection, will receive continued chemotherapy (Arm1, FOLFIRINOX; Arm2, GOFL) 3-4 weeks after CCRT complete. The regimen will continue till disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the exocrine pancreas.
2. Patients must have locally advanced pancreatic cancer (LAPC).
3. Patients must have LAPC evaluated by radiologist and/or surgeon according to either abdominal CT or MRI, or intra-operative findings.

   * Locally advanced unresectable disease was defined by CT or MRI images as low-density tumor (primary and/or lymphadenopathy) with

     1. extension to the celiac axis or superior mesenteric artery,
     2. occlusion of the superior mesenteric-portal venous confluence
     3. aortic, inferior vena cava (IVC) invasion or encasement
     4. invasion of SMV below transverse mesocolon or unresectable after surgical exploration.

   Those who had superior mesenteric vein impingement, superior mesenteric artery abutment were defined as borderline resectable.

   Those who had superior mesenteric vein occlusion, superior mesenteric artery encasement were defined as unresectable.
4. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See section 8.2 for the evaluation of measurable disease.
5. Age >20 years and ≦70 years.
6. ECOG performance score of 0 or 1; see Appendix A.
7. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count >1,500/mL
   * platelets >100,000/mL
   * total bilirubin <1.5X institutional upper limit of normal
   * ALT(SGPT) <5 X institutional upper limit of normal
   * creatinine within normal institutional limits or creatinine clearance>60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
8. Patients who present with jaundice will be allowed to enroll after control with temporary or permanent internal/external drainage.
9. The effects of study agents on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with distant metastases are not eligible.
2. Patients with endocrine or acinar pancreatic carcinoma.
3. Patients may be receiving any steroid, immunologic or other investigational agents within 4 weeks prior to enrollment.
4. Patients who have had prior chemotherapy or radiotherapy are not eligible.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents used in the study.
6. Patients who have above grade II peripheral neuropathy.
7. Patients who had non-curable second primary malignancy within five years, except for non-melanoma skin cancer.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Pregnant women are excluded from this study because the study agents has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated with the study agents.
10. Those who are immuno-compromised or receiving immuno-suppressive therapy are excluded from the study because of increased risk of lethal infections and possible pharmacokinetic interactions with study agent administered during the study.
11. Those who have chronic diarrhea.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
the response rate, disease control rate, overall survival, and patients' quality of life. | 4.5 years
  This is a randomized phase II trial of ICT followed by CCRT with radiotherapy in LAPC. The efficacy will be primarily measured by progression free survival (PFS) as defined in Section 8.5.Other measurements include the response rate, disease control rate, overall survival, and patients' quality of life as described in Section 8.We anticipate that the attrition rate is about 10%, hence, roughly 86 patients will be recruited , we anticipate that the recruitment will be completed in 4.5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Shen, M.D., Principal Investigator — National Cheng-Kung University Hospital; Chih-Hung Hsu, Ph.D., Principal Investigator — National Taiwan University Hospital; Ruey-Kuen Hsieh, M.D., Principal Investigator — Mackay Memorial Hospital; Jen-Shi Chen, M.D., Principal Investigator — Chang Gung Memorial Hospital

REFERENCES:
- [Derived] Su YY, Chiu YF, Li CP, Yang SH, Lin J, Lin SJ, Chang PY, Chiang NJ, Shan YS, Ch'ang HJ, Chen LT. A phase II randomised trial of induction chemotherapy followed by concurrent chemoradiotherapy in locally advanced pancreatic cancer: the Taiwan Cooperative Oncology Group T2212 study. Br J Cancer. 2022 Apr;126(7):1018-1026. doi: 10.1038/s41416-021-01649-7. Epub 2021 Dec 17. PMID 34921230